CLINICAL TRIAL: NCT03578328
Title: TaIwan Network of Targeted Temperature ManagEment for CARDiac Arrest Registry
Brief Title: TaIwan Network of Targeted Temperature ManagEment for CARDiac Arrest Registry (TIMECARD)
Acronym: TIMECARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other); Mackay Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taichung Veterans General Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Changhua Christian Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708013RIND
Record Dates: First submitted 2018-06-12; First posted 2018-07-06 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Arrest; Targeted Temperature Management; Registry
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac arrest with targeted temperature management
  Interventions: Procedure: targeted temperature management

INTERVENTIONS:
Procedure: targeted temperature management — Temperature control to targeted temperature (32-36C) after return of spontaneous circulation after cardiac arrest and resuscitation

SUMMARY:
The goals of the study are to establish the study cohort and database for out-of-hospital cardiac arrest patients. Indications and factors influencing the application of hypothermia treatment on cardiac arrest patients will be analyzed. The prognostic evaluation modalities under hypothermia treatment will be evaluated for their accuracy and optimal time points. These finding and results could be applied in clinical practice in the future.

DETAILED DESCRIPTION:
The importance of cardiopulmonary resuscitation has been emphasized in recent years. The chance of return of spontaneous circulation improves up to 70%. However, only 20 % of cardiac arrest patients can survive to hospital discharge because of post-cardiac arrest syndrome due to global ischemia-reperfusion injuries in cardiac arrest and resuscitation. Although there are some studies trying to predict the survival outcomes in cardiac arrest, the prediction variables are limited to the pre-arrest variables such as age, pre-morbidities. The impact of these variables on long term outcomes is neither clear nor well-defined. It is found that the chances of survival to discharge are significant different among different hospitals and districts. It implies that the intensive managements and treatment policies could influence the outcomes in cardiac arrest patients. However, the critical procedures or managements have not been systemically studied and remain undefined. Targeted temperature management based on hypothermia treatment changes the post-cardiac arrest care and improves the outcome in cardiac arrest patients. Under hypothermia treatment, the critical time points of evaluating prognosis are changed because of 24 hours maintaining cooling period and 12-18 hours rewarming period. The full neurological recovery cannot be evaluated at 24 hours after return of spontaneous circulation as the suggestion in old days without hypothermia treatment. The optimal time points for evaluating and predicting long term outcomes need to be re-defined. The accuracy of different modalities for outcome prediction also needed to be re-evaluated in the hypothermia treatment era. Early and precise prediction of good recovery and favorable outcomes are very important in determining the further intensive treatment strategies by physicians and family for cardiac arrest patients.

The goals of the study are to establish the study cohort and database for out-of-hospital cardiac arrest patients. Indications and factors influencing the application of hypothermia treatment on cardiac arrest patients will be analyzed. The prognostic evaluation modalities under hypothermia treatment will be evaluated for their accuracy and optimal time points. These finding and results could be applied in clinical practice in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧18
2. Non-traumatic cardiac arrest
3. in- or out-of-hospital cardiac arrest requiring cardiopulmonary resuscitation
4. Comatose, defined as Glasgow Coma Score (motor+eye) < 8 or cannot obey verbal command
5. Within 12 hours of return of spontaneous circulation

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, non-traumatic, in- or out-of-hospital cardiac arrest patients after cardiopulmonary resuscitation with return of spontaneous circulation.
  Comatose, defined as Glasgow Coma Score (motor+eye) < 8 or cannot obey verbal command Receiving targeted temperature management within 12 hours after return of spontaneous circulation
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | within one year
favorable neurological outcome when hospital discharge | within one year
  Cerebral Performance Category less than 3

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hua Huang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Derived] Chang HC, Tsai MS, Kuo LK, Hsu HH, Huang WC, Lai CH, Huang CH. Analysis of possible factors affecting neurologic outcomes of resuscitated cardiac arrest patients with initial non-shockable rhythm after targeted temperature management. J Formos Med Assoc. 2025 Apr 2:S0929-6646(25)00143-3. doi: 10.1016/j.jfma.2025.03.025. Online ahead of print. PMID 40180874